CLINICAL TRIAL: NCT02967822
Title: Etude de Génétique moléculaire du Syndrome de Mayer-Rokitansky-Kuster-Hauser
Brief Title: Molecular Genetic Study of Mayer-Rokitansky-Kuster-Hauser Syndrome
Acronym: MRKH
Status: Recruiting | Type: Observational
Sponsor: Imagine Institute (Other)
Collaborators: Reference center for rare diseases (Rare Gynecologic Diseases) (Unknown)
Responsible Party: Sponsor
Other Study IDs: IMNIS2015-06
Record Dates: First submitted 2016-11-14; First posted 2016-11-18 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Mayer Rokitansky Kuster Hauser Syndrome
MeSH Terms: conditions — Mullerian aplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Blood samples (for patients and healthy relatives)
  * Uterine tissue (for patients who have a surgical intervention during their routine follow-up, and only if samples remain available after routine care analyses).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with MRKH syndrome: Biological samples for patients.
  Inclusion of patients presenting MRKH syndrome, and who are followed in clinical centres participating in the study.
  Interventions: Genetic: Biological samples for patients
- Healthy relatives: Biological samples for healthy relatives.
  Inclusion of healthy relatives of patients included in the study (parents, brothers, sisters)
  Interventions: Genetic: Biological samples for healthy relatives

INTERVENTIONS:
Genetic: Biological samples for patients — Blood samples. Sampling of uterine tissue during surgical intervention (collection of samples for the study only if samples remain after the routine care analyses)
  Groups: Patients with MRKH syndrome
Genetic: Biological samples for healthy relatives — Blood samples.
  Groups: Healthy relatives

SUMMARY:
In order to understand the molecular mechanisms leading to Mayer-Rokitansky-Kuster-Hauser syndrome (MRKH), the research team has to identify molecular bases of this anomaly.

Toward this goal, the research team would like to include in the study patients with MRKH syndrome, as well as their healthy relatives, in order to perform genetic analyses, especially whole exome sequencing.

This study has been set up in order to collect biological samples from patients with MRKH and their relatives.

DETAILED DESCRIPTION:
The MRKH is a congenital and rare malformation characterised by the absence of the uterus and of 2/3 of the vagina. The incidence is 1 in 4500 female children (46,XX) and a genetic component has been identified.

In order to understand the molecular mechanisms leading to this disease, the research team has to identify the genetic abnormalities.

This study will be led by the research team of the Imagine Institute and the clinical teams associated with the Reference Center for Rare Diseases PGR (Rare Gynecologic Diseases). Both groups are based on the Necker Hospital campus, and already closely collaborate on research into MRKH syndrome.

This collaboration will allow to :

i) collect biological samples from the propositus and their relatives,

ii) have a medical expertise.

The clinicians involved in the study will recruit patients, whose participation will involve providing a biological sample, ie, a blood sample and/or uterine tissue collected during surgical ablation, in the event that surgery is performed during clinical follow-up of the patients. No specific intervention will be planned for the purposes of this study.

In order to perform genetic analysis on trios, the healthy relatives of the patients (parents, brothers, sisters) will also be included. Blood samples will be taken once for healthy relatives.

Genetic analysis, especially whole exome sequencing, will be performed on blood samples by the research team of Imagine Institute.

ELIGIBILITY:
Inclusion Criteria:

* Patient with MRKH syndrome OR healthy relative of patient included
* Having signed the Informed consent form (or parents in case of patient under 18 years)

Exclusion Criteria:

* Refusal to participate in genetic analyses
* Participation in a therapeutical clinical study in the 30 days prior to inclusion in the present study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Recruitment of patients presenting MRKH syndrome, as well as their healthy relatives, in order to perform genetic analyses
Sampling Method: Probability Sample
Enrollment: 410 (Estimated)
Dates: Start 2016-05; Primary Completion 2031-05 (Estimated); Study Completion 2031-05 (Estimated)

PRIMARY OUTCOMES:
Number of identified nucleotidic variation(s) whose consequences can explain the phenotype of MRKH syndrome | 15 years
  Genetic cause identification

CONTACTS AND LOCATIONS:
Overall Officials: Stanislas Lyonnet, Study Director — Institut Imagine; Michel Polak, Principal Investigator — Necker - Enfants malades hospital
Locations (2):
- France (2):
  - Necker - Enfants malades hospital, Paris
  - Institut Mutualiste Montsouris, Paris

IPD SHARING:
Plan to Share IPD: No